CLINICAL TRIAL: NCT04489498
Title: Comparison of Somatometric Characteristics Between Cerebral Palsy and Normal Children, Cross-sectional, Multi Center Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Other Study IDs: B-1909/562-302
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with stiff cerebral palsy: Children with stiff cerebral palsy, aged 1 to 13 years
- Normal children: Normal children, aged 1 to 13 years

SUMMARY:
The purpose of this study is to: 1) secure basic data of patients with cerebral palsy, 2) seek ways to simplify the data for clinical application, 3) progress of hip dislocation, presence or absence of hip surgery, and The purpose of this study is to compare differences in body development according to severity and nutritional methods.

ELIGIBILITY:
Inclusion Criteria:

* aged 1 to 13
* Experiment group: Children with cerebral palsy, Control group: Normal children
* Patients who agreed to participate in the study

Exclusion Criteria:

* do not agree with the study
* Those who find it difficult to participate under the judgment of the research director

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: It is difficult to find the basis for calculation because there are no papers that measure the body size of children with cerebral palsy and papers that compare with normal children. In particular, children with cerebral palsy are rare diseases, and it is difficult to recruit a large number of subjects.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Anthropometric data (body length) | through study completion, an average of 1 year
  Measure the body length using a tape measure.(cm)
Anthropometric data (BMI) | through study completion, an average of 1 year
  weight and height will be combined to report BMI in kg/m^2
Anthropometric data (body circumference ) | through study completion, an average of 1 year
  Measure the body circumference using a tape measure.(cm)

SECONDARY OUTCOMES:
Progression of hip dislocation | Use simple x-ray within 1 year prior to participation
  It is measured by migration index, which measures the proportion of femoral heads not covered by acetabulum
Progression of scoliosis | Use simple x-ray within 1 year prior to participation
  The degree of scoliosis is measured by Cobbs angle
Have hip dislocation surgery | through study completion, an average of 1 year
  Confirmation of hip dislocation surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Bundang-gu, South Korea